CLINICAL TRIAL: NCT03254485
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study Evaluating the Safety and Efficacy of Different Doses of IW-1973 Over 12 Weeks in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: A Study of the Effect of IW-1973 on the Exercise Capacity of Patients With Heart Failure With Preserved Ejection Fraction (HFpEF)
Acronym: CAPACITY-HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Collaborators: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1973-204
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Cardiovascular; HF; HFpEF
MeSH Terms: conditions — Heart Failure | interventions — praliciguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IW-1973 High Dose (Experimental)
  Interventions: Drug: IW-1973
- Placebo (Placebo Comparator): Placebo to match experimental drug
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: IW-1973 — Oral Tablet
  Arms: IW-1973 High Dose
Drug: Placebo Oral Tablet — Oral Tablet
  Arms: Placebo

SUMMARY:
The objective of the CAPACITY-HFpEF study is to evaluate the safety and efficacy of IW-1973 compared with placebo when administered daily for approximately 12 weeks to patients with HFpEF. The study will evaluate the effect of oral IW-1973 on peak exercise capacity in patients with HFpEF, with or without permanent or persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an ambulatory male or female ≥45 years old at the Screening Visit
2. Patient has heart failure with ejection fraction (EF) of ≥40%
3. Patient has a peak VO2 measuring <80% of age- and sex-adjusted normal values
4. Patient has evidence in medical history supporting clinical heart failure syndrome consisting of at least 1 of the following:

   1. Hospitalization or emergency department visit for heart failure within the past year
   2. Elevated B-type natriuretic peptide (BNP) or N-terminal pro b-type natriuretic peptide (NT-proBNP) within the past 6 months
   3. Echocardiographic evidence within the past 12 months of at least 2 of the following: left ventricular (LV) hypertrophy, left atrial (LA) enlargement, or diastolic dysfunction
   4. Hemodynamic evidence of elevated filling pressures
5. Patient meets at least 2 of the following criteria at the Screening Visit:

   1. Diagnosis of type 2 diabetes mellitus or prediabetes
   2. History of hypertension
   3. Body mass index (BMI) >30 kg/m2
   4. Age ≥70 years

Exclusion Criteria:

1. Patient has had acute coronary syndrome or percutaneous coronary intervention within 30 days before Randomization
2. Patient has had cardiac transplantation or has cardiac transplantation planned during the study
3. Patient has had cardiac artery bypass graft, cardiac mechanical support implantation, or other cardiac surgery in the 3 months before the Screening Visit or planned during the study
4. Patient has severe chronic obstructive coronary disease as defined by chronic oxygen dependence
5. Patient had had heart failure hospitalization with discharge within 30 days before the Screening Visit
6. Patient has a history of clinically significant hypersensitivity or allergies to any of the inactive ingredients contained in the active or placebo drug products
7. Patient has previously received IW-1973 in a study, or received an investigational drug during the 30 days or 5 half lives of that investigational drug (whichever is longer) before the Screening Visit, or is planning to receive another investigational drug at any time during the study
8. Patient is taking specific inhibitors of phosphodiesterase 5 (PDE5), nonspecific inhibitors of PDE5, any supplements for the treatment of erectile dysfunction, riociguat, or nitrates or nitric oxide (NO) donors in any form
9. Patient is taking strong cytochrome P450 3A (CYP3A) inhibitors
10. Women of childbearing potential must have a negative pregnancy test prior to randomization and must agree to use protocol-specified contraception from the Screening Visit through 60 days after the final dose of study drug
11. Male patients must be surgically sterile by vasectomy (conducted ≥60 days before the Screening Visit or confirmed via sperm analysis) or must agree to use protocol-specified contraception from the Screening Visit through 60 days after the final dose of study drug
12. Other exclusion criteria per protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Seferovic, MD PhD, Study Director — Cyclerion Therapeutics, Inc.
Locations (62):
- United States (57):
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - JEHM, La Mesa, California
  - Axis Clinical Trials, Los Angeles, California
  - JEHM, National City, California
  - Valley Clinical Trials, Northridge, California
  - Stanford University, Palo Alto, California
  - Harbor UCLA Medical Center, Torrance, California
  - Aurora Denver Cardiology, Denver, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - PCRS Network, LLC, Miami, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Unity Point Health - Methodist Hospital, Peoria, Illinois
  - Franciscan Physician Network - Indiana Heart Physicians, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lousiana Heart Center, Bogalusa, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Michigan Heart, Ypsilanti, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - VA Healthcare John Cochran Medical Center, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center (OSUMC), Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - PeaceHealth, Sacred Heart Physicians, Springfield, Oregon
  - Research Institute of Lancaster General Health, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North Dallas Research Associates, Dallas, Texas
  - Texas Health Research and Education Insitute, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Schnitzler Cardiovascular Consultants, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University Medical College of Virginia, Richmond, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - Unity Point Health, Madison, Wisconsin
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (5):
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Udelson JE, Lewis GD, Shah SJ, Zile MR, Redfield MM, Burnett J Jr, Parker J, Seferovic JP, Wilson P, Mittleman RS, Profy AT, Konstam MA. Effect of Praliciguat on Peak Rate of Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction: The CAPACITY HFpEF Randomized Clinical Trial. JAMA. 2020 Oct 20;324(15):1522-1531. doi: 10.1001/jama.2020.16641. PMID 33079154
- [Derived] Udelson JE, Lewis GD, Shah SJ, Zile MR, Redfield MM, Burnett J Jr, Mittleman RS, Profy AT, Seferovic JP, Reasner D, Konstam MA. Rationale and design for a multicenter, randomized, double-blind, placebo-controlled, phase 2 study evaluating the safety and efficacy of the soluble guanylate cyclase stimulator praliciguat over 12 weeks in patients with heart failure with preserved ejection fraction (CAPACITY HFpEF). Am Heart J. 2020 Apr;222:183-190. doi: 10.1016/j.ahj.2020.01.009. Epub 2020 Jan 21. PMID 32105984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of different doses of praliciguat (IW-1973) compared with placebo in participants with heart failure with preserved ejection fraction (HFpEF).
Pre-assignment Details: A total of 196 participants were enrolled in the study. Participants enrolled under protocol amendment 2 (or earlier) were randomized in a 1:1:1:1 ratio to 10 milligrams (mg) praliciguat, 20 mg praliciguat, 40 mg praliciguat, or placebo. Participants enrolled under protocol amendment 3 were randomized in a 1:1 ratio to either 40 mg praliciguat or placebo.
Groups:
- Placebo: Participants were randomized to receive matching placebo orally for 12 weeks: 2 weeks of twice daily (BID) dosing followed by 10 weeks of once daily (QD) dosing.
- Praliciguat 10 mg: Participants were randomized to receive praliciguat 10 mg orally for 12 weeks: 2 weeks of BID dosing followed by 10 weeks of QD dosing.
- Praliciguat 20 mg: Participants were randomized to receive praliciguat 20 mg orally for 12 weeks: 2 weeks of BID dosing followed by 10 weeks of QD dosing.
- Praliciguat 40 mg: Participants were randomized to receive praliciguat 40 mg orally for 12 weeks: 2 weeks of BID dosing followed by 10 weeks of QD dosing.
Period: Overall Study
Arm/Group | Placebo | Praliciguat 10 mg | Praliciguat 20 mg | Praliciguat 40 mg
Started | 90 | 7 | 7 | 92
Completed | 78 | 7 | 7 | 77
Not Completed | 12 | 0 | 0 | 15
Not completed — Adverse Event | 3 | 0 | 0 | 6
Not completed — Protocol Violation | 6 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population: The ITT Population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Praliciguat 10 mg | Praliciguat 20 mg | Praliciguat 40 mg | Total
Number analyzed (Participants) | 90 | 7 | 7 | 92 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.0) | 67.3 (9.6) | 69.1 (4.6) | 70.8 (9.1) | 70.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 5 | 3 | 35 | 83
  Male | 50 | 2 | 4 | 57 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 0 | 0 | 20 | 40
  Not Hispanic or Latino | 69 | 7 | 7 | 72 | 155
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 19 | 1 | 2 | 17 | 39
  White | 65 | 6 | 5 | 72 | 148
  More than one race | 2 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Study Drug-related TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as those adverse events (AEs) that started or worsened in severity after the administration of study drug. Causality relationship to study drug was per Investigator assessment. Number of participants with TEAEs and study drug-related TEAEs is presented.
Time Frame: Day 1 up to Day 113
Population: Safety Population consisted of all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Praliciguat 10 mg | Praliciguat 20 mg | Praliciguat 40 mg
Number analyzed (Participants) | 90 | 7 | 7 | 91
Participants
  TEAEs | 61 | 4 | 6 | 72
  Study drug-related TEAEs | 9 | 1 | 0 | 22

2. Primary Outcome: Change From Baseline in Peak Oxygen Consumption (VO2) at Week 12
Description: Peak VO2 was obtained from Cardiopulmonary Exercise Test (CPET), which was used to evaluate the effect of praliciguat on peak exercise capacity. Baseline is defined as the last non-missing measurement prior to the first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the Week 12 value. Data were analyzed using an analysis of covariance (ANCOVA) model with treatment group and atrial fibrillation stratification factors as categorical variable terms and Baseline peak VO2 value as a covariate. Milliliter O2 per kilogram per minute = mL O2/kg/min
Time Frame: Baseline and Week 12
Population: Evaluable Population consisted of all participants in the modified (m)ITT population who completed 8 weeks of dosing (±3 days) and had at least 1 evaluable post-Baseline assessment and did not have a dose reduction. Only those participants with data available at the specified data points were analyzed. Following protocol amendment 3, efficacy analyses included only the praliciguat 40 mg and placebo groups; the praliciguat 10 mg and 20 mg groups were excluded from all efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL O2/kg/min
Arm/Group | Placebo | Praliciguat 40 mg
Number analyzed (Participants) | 72 | 64
mL O2/kg/min | 0.04 [-0.49 to 0.56] | -0.26 [-0.83 to 0.31]
Statistical Analysis 1: Comparison: Placebo vs Praliciguat 40 mg; Test type: Superiority; p = 0.3681, ANCOVA; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.95 to 0.35]

3. Secondary Outcome: Change From Baseline in 6-minute Walk Test (6MWT) Distance at Week 12
Description: 6MWT was a simple assessment of everyday functional capacity and provided a global evaluation of the organ/physiologic systems involved in exercise. 6MWT assessed the distance travelled in 6 minutes, measured at approximately the same time of day. Baseline is defined as the last non-missing measurement prior to the first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the Week 12 value. Data were analyzed using an ANCOVA model with treatment group, atrial fibrillation stratification factor and peak VO2 stratification factor as categorical variable terms and Baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: Evaluable Population. Only those participants with data available at the specified data points were analyzed. Following protocol amendment 3, efficacy analyses included only the praliciguat 40 mg and placebo groups; the praliciguat 10 mg and 20 mg groups were excluded from all efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | Placebo | Praliciguat 40 mg
Number analyzed (Participants) | 72 | 63
Meters | 58.12 [26.12 to 90.11] | 41.38 [8.25 to 74.50]
Statistical Analysis 1: Comparison: Placebo vs Praliciguat 40 mg; Test type: Superiority; p = 0.2817, ANCOVA; Least Squares Mean Difference = -16.74, 95% CI 2-sided [-47.38 to 13.90]

4. Secondary Outcome: Change From Baseline in Ventilatory Efficiency at Week 12
Description: Ventilatory efficiency was defined as minute ventilation/carbon dioxide (VE/VCO2) slope, production and was obtained from CPET. Baseline is defined as the last non-missing measurement prior to the first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the Week 12 value. Data were analyzed using an ANCOVA model with treatment group, atrial fibrillation stratification factor and peak VO2 stratification factor as categorical variable terms and baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: VE/VCO2 Slope
Arm/Group | Placebo | Praliciguat 40 mg
Number analyzed (Participants) | 72 | 64
VE/VCO2 Slope | 0.564 [-0.780 to 1.908] | 0.267 [-1.118 to 1.652]
Statistical Analysis 1: Comparison: Placebo vs Praliciguat 40 mg; Test type: Superiority; p = 0.6508, ANCOVA; Least Squares Mean Difference = -0.297, 95% CI 2-sided [-1.591 to 0.997]

5. Secondary Outcome: CPET Responders at Week 12
Description: CPET responders were defined as participants who improved by at least 1.5 mL O2/kg/min in peak VO2 from Baseline to Week 12. Baseline is defined as the last non-missing measurement prior to the first dose of study drug.
Time Frame: At Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Praliciguat 40 mg
Number analyzed (Participants) | 78 | 65
Participants | 17 | 13

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to Follow-up Visit (Day 113)
Description: TEAEs, defined as those AEs that started or worsened in severity after the initiation of study drug administration are reported for the Safety Population which consisted of all randomized participants who took at least 1 dose of study drug.
Arm/Group | Placebo | Praliciguat 10 mg | Praliciguat 20 mg | Praliciguat 40 mg
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/7 | 0/7 | 1/91
Serious Adverse Events (participants affected / at risk) | 9/90 | 0/7 | 0/7 | 10/91
Other Adverse Events (participants affected / at risk) | 58/90 | 4/7 | 6/7 | 68/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=90) | Praliciguat 10 mg (N=7) | Praliciguat 20 mg (N=7) | Praliciguat 40 mg (N=91)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=90) | Praliciguat 10 mg (N=7) | Praliciguat 20 mg (N=7) | Praliciguat 40 mg (N=91)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1) | 0 (0) | 5 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Therapeutic response unexpected (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 7 (8)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Globulins decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transferrin saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Venous pressure jugular increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 1 (1) | 0 (0) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (9)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pica (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Arterioenteric fistula (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to changes in study objectives and design (protocol amendment 3), all efficacy analyses was performed using only the praliciguat 40 mg and placebo groups; the praliciguat 10 mg and 20 mg groups were excluded from all efficacy analysis. For completeness, participants treated with both 10 mg and 20 mg praliciguat are included in the AE summaries for safety analyses, as well as for Participant Flow and Baseline Characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03254485/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03254485/SAP_001.pdf